CLINICAL TRIAL: NCT02585154
Title: Studying Movement Control in Parkinson's Disease Using Closed Loop Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 168287
Record Dates: First submitted 2015-10-08; First posted 2015-10-23 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: blinded cross-over study of no deep brain stimulation, conventional deep brain stimulation and adaptive deep brain stimulation
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded video assessment

ARMS (3):
- Closed-loop Deep Brain Stimulation (Experimental): Closed-loop Deep Brain Stimulation
  Interventions: Procedure: closed-loop Deep Brain Stimulation applied through custom built external stimulator (Little et al., 2013, 2015); Device: local field potentials and electroencephalography recordings
- Open loop Deep Brain stimulation (Active Comparator): Open loop Deep Brain stimulation
  Interventions: Procedure: Deep Brain Stimulation applied through custom built external stimulator (Little et al., 2013, 2015); Device: local field potentials and electroencephalography recordings
- No Deep Brain Stimulation (Other): No Deep Brain Stimulation
  Interventions: Procedure: Deep Brain Stimulation off; Device: local field potentials and electroencephalography recordings

INTERVENTIONS:
Procedure: Deep Brain Stimulation applied through custom built external stimulator (Little et al., 2013, 2015) — 'Classical' high-frequency Deep Brain Stimulation, which is applied irrespective of ongoing brain activity.
  Arms: Open loop Deep Brain stimulation
Procedure: closed-loop Deep Brain Stimulation applied through custom built external stimulator (Little et al., 2013, 2015) — Deep Brain Stimulation, which is applied depending on ongoing brain activity.
  Arms: Closed-loop Deep Brain Stimulation
Procedure: Deep Brain Stimulation off — Deep Brain Stimulation is turned off.
  Arms: No Deep Brain Stimulation
Device: local field potentials and electroencephalography recordings — Simultaneous recordings of local field potentials from subthalamic nucleus and electroencephalography

SUMMARY:
Parkinson's disease is a common, disabling, progressive condition characterised by severe problems with movement for which medical treatment in the longer term can be unsatisfactory. Deep brain stimulation is a treatment, which directly stimulates the nerve cells affected inside the brain to help overcome the difficulties with movement. Classically, deep brain stimulation stimulates in a manner that is constant and independent of a patients underlying condition as reflected in their brainwave activity. Recent research has suggested that adjusting deep brain stimulation in real time using analyses of brain signals recorded from deep brain stimulation electrodes (termed closed loop deep brain stimulation) nay be better than classical deep brain stimulation in alleviating difficulties with movement. However, it remains unclear whether closed-loop deep brain stimulation also leads to fewer unwanted side effects on movement control. In order to answer this question, the investigators will analyze deep brain stimulation activity and activity recorded from the surface of the head in Parkinson's disease patients undergoing deep brain stimulation surgery. During the recordings patients will perform different movement tasks. Deep brain stimulation has been found to reduce patients' ability to suppress inappropriate movements in certain tasks and performance in these tasks will be the core point of interest. The recordings will be conducted three times: During closed loop deep brain stimulation, classical deep brain stimulation and while the stimulator is turned off. This will allow the investigators to assess putative differences in the effect of closed loop and classical deep brain stimulation with regards to wanted and unwanted effects on movement control and to elucidate their correlates in the brain.

DETAILED DESCRIPTION:
Study Summary Patients will undergo standard 2 part deep brain stimulation implantation (electrode implantation day 1, battery and stimulator implantation approximately day 7, home approximately day 10). The experiments will be performed whilst the patients are inpatients between the two operations and will therefore not require any extra visits or delay in starting therapeutic deep brain stimulation. This paradigm is the standard method for conducting local field potential research in human and represents the paradigm by which the vast majority of previous research in this area has been conducted. Patients will be tested either at Oxford University Hospitals National Health Service Trust or University College London National Health Service Trust.

At least 24h after electrode implantation (first of the two surgeries) patients will be approached about the study and left with the patient information sheet for 24 hours, before further discussion, and, if appropriate consent.

Thereafter, the following procedures will be undertaken:

1. The subjects will participate in a short assessment testing their cognitive function and fill out questionnaires regarding handedness and impulsiveness traits . Furthermore, they will be introduced to the three motor tasks, which they will perform during the definitive test. Together, these assessments will take approximately one hour.

   Prior to the next steps, which will be conducted on the same day or 1-3 days later(depending on the preferences of the participant), participants will be requested to withhold their usual medication overnight so that they are assessed off medication on the morning of the tests.
2. Deep brain stimulation will be evaluated in order to find the best stimulation parameters ( the settings, which yield the best clinical benefit) for each individual patient. This will take approximately 1 hour and is part of the standard clinical procedure.
3. Recordings will be made from the deep brain stimulation electrodes and electrodes placed on the surface of the head in order to assess activity and communication within the brain. During the recordings participants will perform three motor tasks using their hands. In the first two tasks they have to decide whether to press a button on a computer mouse or refrain from a response depending on the nature of some small dots moving in different directions on a computer screen. This will allow assessing patients' ability to perform and inhibit movements. In the third task they are asked to press a button depending on the direction of an arrow presented in the middle of the screen, while ignoring arrows around this central cue. This additional task will allow assessing patients' ability to control conflicting response tendencies. The recordings will be conducted three times: During closed loop deep brain stimulation, open loop deep brain stimulation and while the stimulator is turned off. The order of these sessions will be randomized and counter-balanced across participants. The experimental recordings will take approximately 2 hours.

Prior to recordings we will assess motor impairment using a validated clinical score and patients will have the opportunity to familiarize themselves with the motor tasks.

Completion of the recordings will mark the end of an individual's participation in the study. Given the overall duration of the study patients will be offered the opportunity to complete the recordings after overnight withdrawal of dopaminergic medication over two days or on one single day if preferred.

Thereafter the patient will have their stimulator implanted as usual (most often 7 days after the first operation) and they will be discharged on day 9 - 10 according to their clinical recovery.

For patients with already implanted pacemakers, suitable participants will be identified by the Functional Neurosurgery team who follow the clinical care of the patients. The invitation letter and information sheet will be provided by the clinical team on behalf of the researchers. If patients are interested, they would then be asked to contact the researchers. The same assessments as above (rating scales, motor tasks) will be conducted on one single day in the National Hospital for Neurology and Neurosurgery, London.

Clinical intervention:

Externalisation of electrode wires. The externalisation of the electrode wires will be performed by trained neurosurgeons. This will occur in the awake patient under local anaesthetic (or under a brief general anaesthetic if independent assessment of the patient's clinical state by an anaesthetist determines this to be necessary) in the neurosurgical department.

Research intervention:

Single blinded counterbalanced within-subject trial. Patients will undergo closed loop deep brain stimulation, open loop deep brain stimulation and a session without deep brain stimulation whilst performing motor tasks. Local field potential and electroencephalographic activity will be simultaneously recorded.

Closed loop deep brain stimulation will be delivered through a portable battery operated electronic device connected to the externalised leads. This incorporates an amplifier that allows brain waves to be recorded during deep brain stimulation, a controller and a stimulator. The controller is a simple rectifier and level detector, which then operates a switch that allows stimulation. The level detector is adjusted so that deep brain stimulation is only allowed when a certain clinician determined threshold of pathological brain wave activity is exceeded. The stimulator supplies stimulation at a frequency of 130 Hertz and a voltage as used for standard clinical stimulation. The device weighs about 350 grams and is most simply carried in a small shoulder bag, or attached to a belt.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be Parkinson's disease patients undergoing deep brain stimulation of the subthalamic nucleus (STN).

  * Whether or not a patient is selected for deep brain stimulation surgery is determined by the patient's clinical team purely on independent clinical grounds.
  * Only those patients who have been accepted for deep brain stimulation treatment by their clinical neurologist and functional neurosurgeon will be introduced to the project and have their details passed on to the research team for further information and formal consenting.
* Able to give informed consent.

Exclusion Criteria:

* Lack of capacity to consent (judged by the clinician taking consent as not having sufficient mental capacity to understand the study and its requirements). This is including anyone who, in the opinion of the clinician taking consent, is unlikely to retain sufficient mental capacity for the duration of their involvement in the study.
* Cognitive impairment/lack of capacity to perform experimental task.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ability to suppress inappropriate movements as measured by motor tasks (accuracy measured in %) | Outcome will be assessed on day of experimental sessions (interventions), i.e. the time frame corresponds to the study duration.
Ability to suppress inappropriate movements as measured by motor tasks (response time measured in s) | Outcome will be assessed on day of experimental sessions (interventions), i.e. the time frame corresponds to the study duration.

SECONDARY OUTCOMES:
Local field potential spectra during open-loop deep brain stimulation, closed-loop deep brain stimulation and no deep brain stimulation | Outcome will be assessed on day of experimental sessions (interventions), i.e. the time frame corresponds to the study duration.
  Estimate frequencies from 2 to 35 Hz.
Connectivity between neural regions during open-loop deep brain stimulation, closed-loop deep brain stimulation and no deep brain stimulation | Outcome will be assessed on day of experimental sessions (interventions), i.e. the time frame corresponds to the study duration.
  Estimate frequencies from 2 to 35 Hz.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University College London Hospitals NHS Trust, London
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Background] Little S, Pogosyan A, Neal S, Zavala B, Zrinzo L, Hariz M, Foltynie T, Limousin P, Ashkan K, FitzGerald J, Green AL, Aziz TZ, Brown P. Adaptive deep brain stimulation in advanced Parkinson disease. Ann Neurol. 2013 Sep;74(3):449-57. doi: 10.1002/ana.23951. Epub 2013 Jul 12. PMID 23852650
- [Background] Little S, Beudel M, Zrinzo L, Foltynie T, Limousin P, Hariz M, Neal S, Cheeran B, Cagnan H, Gratwicke J, Aziz TZ, Pogosyan A, Brown P. Bilateral adaptive deep brain stimulation is effective in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2016 Jul;87(7):717-21. doi: 10.1136/jnnp-2015-310972. Epub 2015 Sep 30. PMID 26424898